CLINICAL TRIAL: NCT05169099
Title: Comparative Study of the Results of Trapeziometacarpal Prostheses According to the Preoperative Deformation
Brief Title: Post-operative Results of the Trapezometacarpal (TMC) Prosthesis for Advanced Pre-operative Deformities
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0628
Record Dates: First submitted 2021-11-01; First posted 2021-12-23 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Rhizarthrosis; Arthritis
Keywords: Trapezometacarpal joint arthritis; Adduction angle <25 degrees; Decrease of the grasping and pinching forces; Z deformity of the thumb
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Trapezometacarpal protheses are implanted for patients with trapezometacarpal arthritis. Having a pre-operative thumb adduction angle of less than 25 degrees with hyperextension, meaning a " Z-deformity " are somehow a reason to go for another surgical treatment: trapezectomy with ligament reconstruction. This study will aim at analyzing the results of another surgical treatment which is the trapezometacarpal arthroplasty in this type of deformities.

ELIGIBILITY:
Inclusion criteria:

* Patient with TMC joint arthritis
* Patient with adduction <25 degrees
* Patients with Z deformity
* Patient operated for TMC joint arthroplasty

Exclusion criteria:

- TMC arthroplasty implanted for fractures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated with trapezometacarpal joint arthroplasty for trapezometacarpal joint arthritis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Mobility of the trapezometacarpal joint | 1 day
  Mobility of the trapezometacarpal joint

SECONDARY OUTCOMES:
Number of Participants with Grasping force measured | 1 day
  Grasping force measured
Number of Participants with Pinching force | 1 day
  Pinching force

CONTACTS AND LOCATIONS:
Overall Officials: Michel CHAMMAS, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC